CLINICAL TRIAL: NCT05317806
Title: Use of Metformin in Prevention and Treatment of Cardiac Fibrosis in PAI-1 Deficient Population
Brief Title: Metformin Use in Cardiac Fibrosis in PAI-1 Deficiency
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana Hemophilia &Thrombosis Center, Inc. (Other)
Responsible Party: Principal Investigator, Sweta Gupta, Pediatric Hematologist, Indiana Hemophilia &Thrombosis Center, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2O210069
Record Dates: First submitted 2022-03-08; First posted 2022-04-08 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Plasminogen Activator Inhibitor-1 Deficiency; Cardiac Fibrosis
Keywords: PAI-1 deficiency; Amish; cardiac fibrosis; Metformin
MeSH Terms: conditions — Plasminogen Activator Inhibitor-1 Deficiency | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The study will have one metformin Treatment group (daily metformin administered) and one Observation group (no study drug administered)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin Treatment Group (Experimental): Subjects with PAI-1 deficiency with or without cardiac fibrosis, receiving daily treatment with metformin for a daily range of 500-2000mg
  Interventions: Drug: Metformin Extended Release Oral Tablet
- Observation Group (No Intervention): Subjects with PAI-1 deficiency with or without cardiac fibrosis, not receiving treatment with metformin
  Subjects are allowed to switch between the two groups

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — daily metformin treatment vs. no treatment with metformin
  Other Names: Glucophage XR
  Arms: Metformin Treatment Group

SUMMARY:
This study will evaluate the efficacy and safety of metformin, in patients 18-65 years of age with homozygous plasminogen activator inhibitor-1 (PAI-1) deficiency, with or without cardiac fibrosis, for a period of 60 months. The starting dose of metformin will be 500 mg up to a maximum dose of 2000 mg for a period of 5 years with the aim to assess the safety and efficacy of metformin on prevention/stabilization or regression of cardiac fibrosis in a Treated population vs. a Comparison population.

DETAILED DESCRIPTION:
This study is a phase 4, prospective, open-label, US single center study to assess the efficacy and safety of metformin for prevention or stabilization or regression of cardiac fibrosis in individuals homozygous for PAI-1 deficiency. Approximately 15 patients 18-65 years of age are expected to be enrolled, due to the rarity of this blood disorder. The study will have one metformin Treatment group (daily metformin administered) and one Observation group (no study drug administered). Subjects will be consented and screened by Indiana Hemophilia and Thrombosis Center (IHTC) staff. Individuals will be eligible for study participation if they meet all inclusion criteria. Subjects will be excluded from the study if they meet any of the exclusion criteria. US-labeled oral metformin (extended release) will be administered using the FDA-approved dosing regimen for diabetes mellitus type II starting at a dose of 500 mg and escalating up to a maximum of 2000 mg. In the final assessment, subjects who receive metformin for at least 36 months (and up to a maximum of 60 months) will be considered part of the Treated population. Subjects who refuse treatment with metformin or complete <36 months of treatment on metformin either due to intolerance to the study drug or due to any other reason, will be considered part of the Comparison population and will be followed clinically. Females will be offered the option to temporarily discontinue metformin during pregnancy and/or lactation period; they will be considered part of the Treated population if they receive metformin for at least 36 months during the study (those 36 months need not be consecutive). If they receive metformin for 0 to <36 months, they will be considered part of the Comparison population. The study enrollment period will be 12 months. Every subject will be in the study for a period of 60 months from the point of enrollment. There is no minimum on-study period. The decision to continue metformin treatment beyond the study period in the metformin Treatment group, will be made based on drug efficacy, patient tolerability/preference, and provider discretion.

Basic laboratory parameters (serum chemistry and hematology), specific cardiac markers (NT-pro BNP, TGF-β1) cardiac imaging and electrocardiograms will be performed at baseline, at study close out/subject withdrawal, and as specified in the schedule of activities. Adverse events (AE) will be recorded on an ongoing basis as they occur during the study. During the study, annual cardiac consultation, New York Heart Association (NYHA) scale and as needed, the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) will be completed by patients.

The primary analysis will be performed when the last patient has completed 60 months in the study, is lost to follow up or has withdrawn from the study treatment, whichever occurs first.

An interim analysis will be performed at 30 months. All patients will be included in the interim analysis. This interim analysis will be performed for safety.

Definitions

• Complete PAI-1 deficiency defined as subjects with homozygous mutation in SERPINE 1.

During the clinical trial, subjects will be grouped according to whether they are currently receiving study drug or not. This will affect the schedule of study visits and assays/procedures performed.

* Metformin Treatment group: The group of individuals who are currently receiving metformin
* Observation group: The group of individuals who are NOT currently receiving metformin (this includes those who opted to never receive metformin) Patients will be allowed to switch between metformin treatment group and observation group.

Following the completion of the clinical trial, subjects will be grouped according to the total amount of time they received study drug. This grouping is for analytical/statistical purposes only.

* Treated population: Individuals who received at least 36 months of metformin treatment while on study
* Comparison population: Individuals who did not receive metformin treatment at any point during the study, or received metformin for a total less than 36 months of treatment while on study i.e. 0 to <36 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Confirmed homozygosity for mutation in SERPINE-1 for PAI-1 deficiency
* Male or female
* Aged 18-65 years
* Willing and able to choose between being in a metformin Treatment group (daily metformin) or an Observation group (no study drug) at study entry
* Capable of understanding and willing to comply with the conditions of the study (in the opinion of the study investigator(s))
* Have read, understood and be able to provide written informed consent

Exclusion Criteria:

* Not homozygous for SERPINE-1 mutation for PAI-1 deficiency, based on genetic testing
* Ages <18 or >65 years
* Renal dysfunction (Cockcroft Gault CrCl < 30)
* History of hypersensitivity of metformin or any component in the extended release formulation
* Unwillingness to avoid alcohol
* Currently prescribed cimetidine, dolutegravir, patiromer, ranolazine, or tafenoquine and no alternate therapy is possible
* History of illicit drug or alcohol abuse within 48 weeks prior to screening, in the study investigators' judgment
* Concomitant disease, condition, significant abnormality on screening evaluations or laboratory tests, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the study investigator(s), pose an additional unacceptable risk in administering study drug to the patient
* Receipt of any other investigational medicinal product currently being administered (or planned to be administered)
* Inability to comply with the study protocol (in the opinion of the study investigator(s))
* Inability to understand and provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of individuals homozygous for PAI-1 deficiency with stable or improved cardiac fibrosis | through the study annually, up to 60 months
  Measured using cardiac MRI to quantify the percentage cardiac fibrosis.
Number of individuals homozygous for PAI-1 deficiency with stable or improved Transforming growth factor (TGF-β1) | through the study annually, up to 60 months
  Measured by a blood draw as a surrogate marker for status of cardiac fibrosis stability or reduction.

SECONDARY OUTCOMES:
Number of individuals homozygous for PAI-1 deficiency with metformin related adverse events as assessed by grading of diarrhea (CTCAE v5.0) | approximately monthly (±4 weeks) until maximum tolerated dose for metformin is achieved until 6 months (±4 weeks) and then every 3 months (±4 weeks) for the entire study period for the metformin group
  Safety and tolerability of metformin when administered to individuals homozygous for PAI-1 deficiency as assessed by side effect profile (as measured by the type and number of adverse drug reactions and serious adverse drug reactions )
Number of individuals homozygous for PAI-1 deficiency with clinical symptoms of heart failure as measured by the New York Heart Association (NYHA) scale and as needed, the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 6 months after study enrollment, through the study annually, up to 60 months
  Objective evaluation of cardiac symptoms by using a scale and questionnaire.
  New York Heart Association (NYHA) scale: lowest scale is Functional capacity I, Objective assessment A; Highest scale is Functional capacity IV, Objective assessment D. Higher scores worst outcome.
Number of individuals homozygous for PAI-1 deficiency with additional signs of heart failure assessed by measuring N- terminal prohormone beta natriuretic peptide (NT-pro BNP) | through the study annually, up to 60 months
  Objective evaluation of heart failure using NT-proBNP value as stable, increasing or decreasing
Number of individuals homozygous for PAI-1 deficiency with stable or improved ejection fraction on echocardiogram | through the study annually, up to 60 months
  Evaluate changes in ejection fraction by standard transthoracic echocardiogram
Number of individuals homozygous for PAI-1 deficiency with clinical symptoms of heart failure impacting their health as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 6 months after study enrollment, through the study annually, up to 60 months
  Objective evaluation of cardiac failure symptoms impact on health by using a questionnaire.
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12): KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent. Higher scores are better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sweta Gupta, MD, Principal Investigator — Indiana Hemophilia and Thrombosis Center, Inc; Magdalena Lewandowska, MD, Principal Investigator — Indiana Hemophilia and Thrombosis Center, Inc; Amy D Shapiro, MD, Study Director — Indiana Hemophilia and Thrombosis Center, Inc
Locations (1):
- Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
TBD based on analysis
Supporting Information: Study Protocol, ICF
Time Frame: Post analysis

REFERENCES:
- [Background] Loskutoff DJ, Sawdey M, Mimuro J. Type 1 plasminogen activator inhibitor. Prog Hemost Thromb. 1989;9:87-115. No abstract available. PMID 2492381
- [Background] Chmielewska J, Ranby M, Wiman B. Evidence for a rapid inhibitor to tissue plasminogen activator in plasma. Thromb Res. 1983 Aug 1;31(3):427-36. doi: 10.1016/0049-3848(83)90407-3. PMID 20217999
- [Background] Chmielewska J, Ranby M, Wiman B. Kinetics of the inhibition of plasminogen activators by the plasminogen-activator inhibitor. Evidence for 'second-site' interactions. Biochem J. 1988 Apr 15;251(2):327-32. doi: 10.1042/bj2510327. PMID 3135797
- [Background] Mehta R, Shapiro AD. Plasminogen activator inhibitor type 1 deficiency. Haemophilia. 2008 Nov;14(6):1255-60. doi: 10.1111/j.1365-2516.2008.01834.x. PMID 19141166
- [Background] Fay WP, Parker AC, Condrey LR, Shapiro AD. Human plasminogen activator inhibitor-1 (PAI-1) deficiency: characterization of a large kindred with a null mutation in the PAI-1 gene. Blood. 1997 Jul 1;90(1):204-8. PMID 9207454
- [Background] Fay WP, Shapiro AD, Shih JL, Schleef RR, Ginsburg D. Brief report: complete deficiency of plasminogen-activator inhibitor type 1 due to a frame-shift mutation. N Engl J Med. 1992 Dec 10;327(24):1729-33. doi: 10.1056/NEJM199212103272406. No abstract available. PMID 1435917
- [Background] Iwaki T, Tanaka A, Miyawaki Y, Suzuki A, Kobayashi T, Takamatsu J, Matsushita T, Umemura K, Urano T, Kojima T, Terao T, Kanayama N. Life-threatening hemorrhage and prolonged wound healing are remarkable phenotypes manifested by complete plasminogen activator inhibitor-1 deficiency in humans. J Thromb Haemost. 2011 Jun;9(6):1200-6. doi: 10.1111/j.1538-7836.2011.04288.x. PMID 21486382
- [Background] Iwaki T, Nagahashi K, Kobayashi T, Umemura K, Terao T, Kanayama N. The first report of uncontrollable subchorionic and retroplacental haemorrhage inducing preterm labour in complete PAI-1 deficiency in a human. Thromb Res. 2012 Apr;129(4):e161-3. doi: 10.1016/j.thromres.2011.10.008. Epub 2011 Nov 17. No abstract available. PMID 22099705
- [Background] Iwaki T, Nagahashi K, Takano K, Suzuki-Inoue K, Kanayama N, Umemura K, Urano T. Mutation in a highly conserved glycine residue in strand 5B of plasminogen activator inhibitor 1 causes polymerisation. Thromb Haemost. 2017 May 3;117(5):860-869. doi: 10.1160/TH16-07-0572. Epub 2017 Feb 23. PMID 28229167
- [Background] Angleton P, Chandler WL, Schmer G. Diurnal variation of tissue-type plasminogen activator and its rapid inhibitor (PAI-1). Circulation. 1989 Jan;79(1):101-6. doi: 10.1161/01.cir.79.1.101. PMID 2491971
- [Background] Heiman M, Gupta S, Shapiro AD. The obstetric, gynaecological and fertility implications of homozygous PAI-1 deficiency: single-centre experience. Haemophilia. 2014 May;20(3):407-12. doi: 10.1111/hae.12313. Epub 2013 Nov 22. PMID 24261743
- [Background] Flevaris P, Vaughan D. The Role of Plasminogen Activator Inhibitor Type-1 in Fibrosis. Semin Thromb Hemost. 2017 Mar;43(2):169-177. doi: 10.1055/s-0036-1586228. Epub 2016 Aug 24. PMID 27556351
- [Background] Ghosh AK, Vaughan DE. PAI-1 in tissue fibrosis. J Cell Physiol. 2012 Feb;227(2):493-507. doi: 10.1002/jcp.22783. PMID 21465481
- [Background] Ghosh AK, Bradham WS, Gleaves LA, De Taeye B, Murphy SB, Covington JW, Vaughan DE. Genetic deficiency of plasminogen activator inhibitor-1 promotes cardiac fibrosis in aged mice: involvement of constitutive transforming growth factor-beta signaling and endothelial-to-mesenchymal transition. Circulation. 2010 Sep 21;122(12):1200-9. doi: 10.1161/CIRCULATIONAHA.110.955245. Epub 2010 Sep 7. PMID 20823384
- [Background] Xu Z, Castellino FJ, Ploplis VA. Plasminogen activator inhibitor-1 (PAI-1) is cardioprotective in mice by maintaining microvascular integrity and cardiac architecture. Blood. 2010 Mar 11;115(10):2038-47. doi: 10.1182/blood-2009-09-244962. Epub 2009 Dec 15. PMID 20009036
- [Background] Khan SS, Shah SJ, Strande JL, Baldridge AS, Flevaris P, Puckelwartz MJ, McNally EM, Rasmussen-Torvik LJ, Lee DC, Carr JC, Benefield BC, Afzal MZ, Heiman M, Gupta S, Shapiro AD, Vaughan DE. Identification of Cardiac Fibrosis in Young Adults With a Homozygous Frameshift Variant in SERPINE1. JAMA Cardiol. 2021 Jul 1;6(7):841-846. doi: 10.1001/jamacardio.2020.6909. PMID 33439236
- [Background] Flevaris P, Khan SS, Eren M, Schuldt AJT, Shah SJ, Lee DC, Gupta S, Shapiro AD, Burridge PW, Ghosh AK, Vaughan DE. Plasminogen Activator Inhibitor Type I Controls Cardiomyocyte Transforming Growth Factor-beta and Cardiac Fibrosis. Circulation. 2017 Aug 15;136(7):664-679. doi: 10.1161/CIRCULATIONAHA.117.028145. Epub 2017 Jun 6. PMID 28588076
- [Background] Joshi N, Kopec AK, Towery K, Williams KJ, Luyendyk JP. The antifibrinolytic drug tranexamic acid reduces liver injury and fibrosis in a mouse model of chronic bile duct injury. J Pharmacol Exp Ther. 2014 Jun;349(3):383-92. doi: 10.1124/jpet.113.210880. Epub 2014 Mar 14. PMID 24633426
- [Background] King P, Peacock I, Donnelly R. The UK prospective diabetes study (UKPDS): clinical and therapeutic implications for type 2 diabetes. Br J Clin Pharmacol. 1999 Nov;48(5):643-8. doi: 10.1046/j.1365-2125.1999.00092.x. No abstract available. PMID 10594464
- [Background] Sasali A, Leahy JL. Is metformin cardioprotective? Diabetes Care. 2003 Jan;26(1):243-4. doi: 10.2337/diacare.26.1.243. No abstract available. PMID 12502689
- [Background] Choi SM, Jang AH, Kim H, Lee KH, Kim YW. Metformin Reduces Bleomycin-induced Pulmonary Fibrosis in Mice. J Korean Med Sci. 2016 Sep;31(9):1419-25. doi: 10.3346/jkms.2016.31.9.1419. PMID 27510385
- [Background] Kita Y, Takamura T, Misu H, Ota T, Kurita S, Takeshita Y, Uno M, Matsuzawa-Nagata N, Kato K, Ando H, Fujimura A, Hayashi K, Kimura T, Ni Y, Otoda T, Miyamoto K, Zen Y, Nakanuma Y, Kaneko S. Metformin prevents and reverses inflammation in a non-diabetic mouse model of nonalcoholic steatohepatitis. PLoS One. 2012;7(9):e43056. doi: 10.1371/journal.pone.0043056. Epub 2012 Sep 18. PMID 23028442
- [Background] Ursini F, Grembiale RD, D'Antona L, Gallo E, D'Angelo S, Citraro R, Visca P, Olivieri I, De Sarro G, Perrotti N, Russo E. Oral Metformin Ameliorates Bleomycin-Induced Skin Fibrosis. J Invest Dermatol. 2016 Sep;136(9):1892-1894. doi: 10.1016/j.jid.2016.05.097. Epub 2016 May 29. No abstract available. PMID 27251791
- [Background] Wang M, Weng X, Guo J, Chen Z, Jiang G, Liu X. Metformin alleviated EMT and fibrosis after renal ischemia-reperfusion injury in rats. Ren Fail. 2016;38(4):614-21. doi: 10.3109/0886022X.2016.1149770. Epub 2016 Feb 26. PMID 26915376
- [Background] Xiao H, Ma X, Feng W, Fu Y, Lu Z, Xu M, Shen Q, Zhu Y, Zhang Y. Metformin attenuates cardiac fibrosis by inhibiting the TGFbeta1-Smad3 signalling pathway. Cardiovasc Res. 2010 Aug 1;87(3):504-13. doi: 10.1093/cvr/cvq066. Epub 2010 Mar 3. PMID 20200042
- [Background] Xu S, Yang Z, Jin P, Yang X, Li X, Wei X, Wang Y, Long S, Zhang T, Chen G, Sun C, Ma D, Gao Q. Metformin Suppresses Tumor Progression by Inactivating Stromal Fibroblasts in Ovarian Cancer. Mol Cancer Ther. 2018 Jun;17(6):1291-1302. doi: 10.1158/1535-7163.MCT-17-0927. Epub 2018 Mar 15. PMID 29545331
- [Background] McCloskey CW, Cook DP, Kelly BS, Azzi F, Allen CH, Forsyth A, Upham J, Rayner KJ, Gray DA, Boyd RW, Murugkar S, Lo B, Trudel D, Senterman MK, Vanderhyden BC. Metformin Abrogates Age-Associated Ovarian Fibrosis. Clin Cancer Res. 2020 Feb 1;26(3):632-642. doi: 10.1158/1078-0432.CCR-19-0603. Epub 2019 Oct 9. PMID 31597663
- [Background] De Souza A, Khawaja KI, Masud F, Saif MW. Metformin and pancreatic cancer: Is there a role? Cancer Chemother Pharmacol. 2016 Feb;77(2):235-42. doi: 10.1007/s00280-015-2948-8. Epub 2016 Jan 6. PMID 26740120
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Liu Q, Li S, Quan H, Li J. Vitamin B12 status in metformin treated patients: systematic review. PLoS One. 2014 Jun 24;9(6):e100379. doi: 10.1371/journal.pone.0100379. eCollection 2014. PMID 24959880
- [Background] Carrizo E, Fernandez V, Connell L, Sandia I, Prieto D, Mogollon J, Valbuena D, Fernandez I, de Baptista EA, Baptista T. Extended release metformin for metabolic control assistance during prolonged clozapine administration: a 14 week, double-blind, parallel group, placebo-controlled study. Schizophr Res. 2009 Aug;113(1):19-26. doi: 10.1016/j.schres.2009.05.007. Epub 2009 Jun 9. PMID 19515536
- [Background] Rado J, von Ammon Cavanaugh S. A Naturalistic Randomized Placebo-Controlled Trial of Extended-Release Metformin to Prevent Weight Gain Associated With Olanzapine in a US Community-Dwelling Population. J Clin Psychopharmacol. 2016 Apr;36(2):163-8. doi: 10.1097/JCP.0000000000000469. PMID 26872112
- [Background] Lipska KJ, Bailey CJ, Inzucchi SE. Use of metformin in the setting of mild-to-moderate renal insufficiency. Diabetes Care. 2011 Jun;34(6):1431-7. doi: 10.2337/dc10-2361. No abstract available. PMID 21617112
- [Background] Inzucchi SE, Lipska KJ, Mayo H, Bailey CJ, McGuire DK. Metformin in patients with type 2 diabetes and kidney disease: a systematic review. JAMA. 2014 Dec 24-31;312(24):2668-75. doi: 10.1001/jama.2014.15298. PMID 25536258
- [Background] Kilo C. Metformin: a safe and effective treatment in the management of NIDDM. Mo Med. 1997 Mar;94(3):114-23. PMID 9071866
- [Background] Johnson NP. Metformin use in women with polycystic ovary syndrome. Ann Transl Med. 2014 Jun;2(6):56. doi: 10.3978/j.issn.2305-5839.2014.04.15. PMID 25333031
- See also: Gupta S, Sealls W, Shapiro A. Rare coagulation disorders resource room - plasminogen activator inbitor type 1 deficiency. Rare coagulation disorders resource room [cited August 8, 2019] — https://www.rarecoagulationdisorders.org/